CLINICAL TRIAL: NCT04021290
Title: A Phase III, Randomized, Multicenter, Open-label, Non-inferiority Study Evaluating the Efficacy, Safety and Tolerability of Switching to Dolutegravir/Lamivudine Fixed Dose Combination in HIV-1 Infected Adults Who Are Virologically Suppressed
Brief Title: Regimen Switch to Dolutegravir/Lamivudine Fixed Dose Combination From Current Antiretroviral Regimen in HIV-1 Infected and Virologically Suppressed Adults (SALSA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry); PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 208090
Record Dates: First submitted 2019-07-11; First posted 2019-07-16 (Actual); Results first posted 2022-07-01 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: HIV Infections
Keywords: Current antiretroviral regimen (CAR); HIV-1; Long-term antiviral activity; Dolutegravir/lamivudine; Fixed dose combination
MeSH Terms: conditions — HIV Infections | interventions — Automobiles

STUDY DESIGN:
Intervention Model Description: This is a randomized study with parallel group assignment where participants will be randomized into one of the two treatment groups. Participants randomized to DTG/3TC FDC will receive DTG/3TC FDC up to Week 52. Participants randomized to CAR will continue to take their current regimen up to Week 52. Randomization will be stratified by Baseline third agent class (protease inhibitor [PI], integrase inhibitor [INI], or non-nucleoside reverse transcriptase inhibitor [NNRTI]).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants receiving DTG/3TC FDC (Experimental): Eligible participants will be randomized to receive 50 milligrams (mg)/300 mg DTG/3TC FDC therapy from Day 1 up to 52 weeks. Participants who complete 52 weeks of treatment will have the opportunity to continue receiving DTG/3TC FDC once daily in the continuation phase.
  Interventions: Drug: DTG/3TC FDC
- Participants receiving CAR (Active Comparator): Eligible participants will continue to receive CAR from Day 1 up to 52 weeks.
  Interventions: Drug: CAR

INTERVENTIONS:
Drug: DTG/3TC FDC — DTG/3TC FDC will be available as white, oval, film-coated tablets at a unit dose strength of 50 mg/300 mg. Participants will take DTG/3TC once daily via oral route.
  Arms: Participants receiving DTG/3TC FDC
Drug: CAR — Participants who are randomized to the CAR arm will continue to take the current treatment until Week 52. CAR will include 2 NTRIs plus either an INI, NNRTI, or boosted PI or atazanavir unboosted.
  Arms: Participants receiving CAR

SUMMARY:
The aim of this study is to determine if virologically suppressed Human Immunodeficiency Virus (HIV) Type 1 infected adults on a current antiretroviral regimen (CAR) (including 2 nucleoside reverse transcriptase inhibitors [NRTIs] plus a third agent) remain suppressed upon switching to dolutegravir/lamivudine (DTG/3TC) fixed dose combination (FDC). The main objective of the study is to demonstrate the non-inferior antiviral activity of switching to DTG/3TC FDC once daily compared to continuation of CAR over 48 weeks in virologically suppressed adults living with HIV-1. The study will also evaluate information regarding the safety and health related quality of life. The study will include Screening Phase (up to 28 days), a Randomization Phase (up to Week 52) and a Continuation Phase (post Week 52). The Continuation Phase is not applicable for participants in Sweden and Denmark. Approximately 490 participants will be randomized in 1:1 ratio to receive DTG/3TC FDC once daily for up to 52 weeks or continue their CAR for 52 weeks. Participants in the DTG/3TC FDC arm who successfully complete up to 52 weeks of treatment will have the opportunity to continue receiving DTG/3TC FDC once daily in Continuation Phase.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants must be able to understand and comply with protocol requirements, instructions, and restrictions; participant must be likely to complete the study as planned; participants should be considered appropriate candidates for participation in an investigative clinical trial with oral medication (example given [e.g.] no active problematic substance abuse, acute major organ disease, or potential long-term work assignments out of the country).
* Participant should be aged 18 years or older (or older, if required by local regulatory agencies), at the time of signing the informed consent.
* Participants living with HIV.
* Documented evidence of at least two plasma HIV-1 RNA measurements <50 c/mL in the 12 months prior to Screening: one within the 6 to 12 month window, and one within 6 months prior to Screening.
* Plasma HIV-1 RNA <50 c/mL at Screening.
* Participant must be on uninterrupted current regimen (either the initial or second Combination antiretroviral therapy [cART] regimen) for at least 3 months prior to Screening.

  i) Any prior switch, defined as a change of a single drug or multiple drugs simultaneously, must have occurred due to tolerability and/or safety concerns or access to medications, or convenience/simplification and must not have been done for suspected or established treatment failure. The following switches, if they are the only switches, would not be considered a change in regimen. a) A switch from a PI boosted with ritonavir (RTV) to the same PI boosted with cobicistat is allowed (and vice versa). b) A switch from 3TC to emtricitabine (FTC) (and vice versa). c) A switch from tenofovir disoproxil fumarate (TDF) to tenofovir alafenamide (TAF) (and vice versa).

ii) Acceptable stable cART regimens prior to Screening include 2 NRTIs plus a) INI (either the initial or second cART regimen) b) NNRTI (either the initial or second cART regimen) c) Boosted PI (or atazanavir [ATV] unboosted) (either the initial or second PI-based cART regimen).

* A male or female participant.
* A female participant is eligible to participate if she is not pregnant [as confirmed by a negative serum human chorionic gonadotrophin (hCG) test at screen and a negative urine hCG test at randomization (a local serum hCG test at randomization is allowed if it can be done, and results obtained, within 24 hours prior to randomization)], not breastfeeding, and at least one of the following conditions applies; not a woman of childbearing potential (WOCBP) or a WOCBP who agrees to follow the contraceptive guidance during the treatment period from 28 days prior to the first dose of study medication and for at least 2 weeks after the last dose of study medication. All participants in the study should be counseled on safer sexual practices including the use and benefit/risk of effective barrier methods (e.g., male condom) and on the risk of HIV transmission to an uninfected partner; The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Participant must be capable of giving signed informed consent.
* Participants enrolled in France must be affiliated to, or a beneficiary of, a social security category.

Exclusion Criteria:

* Women who are pregnant or breastfeeding or plan to become pregnant or breastfeed during the study.
* Any evidence of an active Centers for Disease Control and Prevention (CDC) Stage 3 disease except cutaneous Kaposi's sarcoma not requiring systemic therapy. Historical or current CD4 cell counts less than 200 cells per cubic millimeter (mm^3) are not exclusionary.
* Participants with severe hepatic impairment (Class C) as determined by Child-Pugh classification.
* Participants with unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Participants with the evidence of Hepatitis B virus (HBV) infection based on the results of testing at Screening for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (anti-HBc), Hepatitis B surface antigen antibody (anti-HBs) and HBV deoxyribonucleic acid (DNA) as follows: Participants positive for HBsAg are excluded; Participants negative for anti-HBs but positive for anti-HBc (negative HBsAg status) and positive for HBV DNA are excluded. Participant's positive for anti-HBc (negative HBsAg status) and positive for anti-HBs (past and/or current evidence) are immune to HBV and are not excluded. Anti-HBc must be either total anti-HBc or anti-HBc immunoglobulin G (IgG), and not anti-HBc Immunoglobulin M (IgM). Participants with a documented history of chronic HBV and current undetectable HBV DNA while on a TAF/TDF regimen are excluded.
* Participants with anticipated need for any hepatitis C virus (HCV) therapy during the randomized phase of the study, or anticipated need for HCV therapy with a potential for adverse drug-drug interactions with DTG or 3TC.
* Participants with untreated syphilis infection (positive rapid plasma reagin [RPR] at Screening without clear documentation of treatment). Participants who are at least 7 days post completed treatment are eligible.
* Participants with history or presence of allergy intolerance to the study interventions or their components or drugs of their class.
* Participants with ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical, anal or penile intraepithelial neoplasia.
* Participants who in the investigator's judgment, poses a significant suicidality risk.
* Participants with any pre-existing physical or mental condition which, in the opinion of the Investigator, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant.
* Any condition which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or excretion of the study interventions or render the participant unable to take oral medication.
* Use of any regimen consisting of single or dual ART (peri-partum treatment with single dose nevirapine is allowed).
* Participants with current use of stavudine, didanosine, or nelfinavir.
* Participants receiving any prohibited medication and who are unwilling or unable to switch to an alternate medication.
* Participants receiving treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening.
* Participants receiving treatment with any of the following agents within 28 days of Screening like radiation therapy; cytotoxic chemotherapeutic agents; any systemic immune suppressant.
* Participants with exposure to an experimental drug or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of investigational product (IP).
* Any evidence of major NRTI mutation or presence of any DTG resistance-associated mutation in any available prior resistance genotype assay test result, if known.
* Participants with any verified Grade 4 laboratory abnormality, with the exception of Grade 4 lipid abnormalities. A single repeat test is allowed during the Screening period to verify a result.
* Participants with alanine aminotransferase (ALT) >= 5 times the upper limit of normal (ULN) or ALT >= 3 times ULN and bilirubin >= 1.5 times ULN (with >35 percent direct bilirubin).
* Participants with creatinine clearance of <30 mL/min/1.73m^2 via Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) method. Participants with creatinine clearance between 30 to 49 mL/min/1.73 m^2 are eligible after the medical monitor has provided approval after reviewing participant's current ART regimen.
* Participants with any acute laboratory abnormality at Screening, which, in the opinion of the investigator, would preclude the participant'sparticipation in the study of an investigational compound.
* Participants within the 12 month window prior to Screening and after confirmed suppression to <50 c/mL, any plasma HIV-1 RNA measurement >200 c/mL.
* Participants within the 12 month window prior to Screening and after confirmed suppression to <50 c/mL, 2 or more consecutive plasma HIV-1 RNA measurements >=50 c/mL. A single plasma HIV-1 RNA measurement >50 c/mL but less than 200 c/mL, with confirmation of return to <50 c/mL is allowed.
* Any history of switch to another regimen, defined as change of a single drug or multiple drugs simultaneously, due to virologic failure to therapy (defined as a confirmed plasma HIV-1 RNA >=400 c/mL).
* Participants with any drug holiday during the 6 months prior to Screening, except for brief periods (less than 1 month) where all ART was stopped due to tolerability and/or safety concerns.
* Participants who are currently participating in or anticipate to be selected for any other interventional study after randomization.
* Participants enrolled in France (or in other countries as required by local regulations or Ethics Committee/Institutional Review Board [IRB]) who participated in any study using an investigational drug or vaccine during the previous 60 days or 5 half-lives, or twice the duration of the biological effect of the experimental drug or vaccine, whichever is longer, prior to screening for the study, or participate simultaneously in another clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2022-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (101):
- United States (15):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Hillsborough, New Jersey
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Morgantown, West Virginia
  - GSK Investigational Site, Milwaukee, Wisconsin
- Argentina (4):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
- Belgium (3):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
- Brazil (6):
  - GSK Investigational Site, Salvador, Estado de Bahia
  - GSK Investigational Site, Curitiba, Paraná
  - GSK Investigational Site, Campinas, São Paulo
  - GSK Investigational Site, Manaus
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, São Paulo
- Canada (6):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Regina, Saskatchewan
- China (4):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Shanghai
- Denmark (4):
  - GSK Investigational Site, Aarhus
  - GSK Investigational Site, Copenhagen
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, Odense C
- France (7):
  - GSK Investigational Site, Bobigny
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Orléans
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Tourcoing
- Germany (8):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, München, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, München
- Italy (6):
  - GSK Investigational Site, Modena, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Bergamo
  - GSK Investigational Site, Brescia
- Mexico (3):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Distrito Federal
- Russia (3):
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Tolyatti
  - GSK Investigational Site, Yekaterinburg
- South Africa (3):
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Observatory, Cape Town
- Spain (11):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Badalona, Barcelona
  - GSK Investigational Site, Cadiz
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, San Sebastián de los Reyes
  - GSK Investigational Site, Santa Cruz de Tenerife
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
- Sweden (3):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Stockholm
- Taiwan (6):
  - GSK Investigational Site, Kaohsiumg
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, New Taipei City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District
- United Kingdom (9):
  - GSK Investigational Site, Leeds, Yorkshire
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Brighton
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Llibre JM, Brites C, Cheng CY, Osiyemi O, Galera C, Hocqueloux L, Maggiolo F, Degen O, Taylor S, Blair E, Man C, Wynne B, Oyee J, Underwood M, Curtis L, Bontempo G, van Wyk J. Efficacy and Safety of Switching to the 2-Drug Regimen Dolutegravir/Lamivudine Versus Continuing a 3- or 4-Drug Regimen for Maintaining Virologic Suppression in Adults Living With Human Immunodeficiency Virus 1 (HIV-1): Week 48 Results From the Phase 3, Noninferiority SALSA Randomized Trial. Clin Infect Dis. 2023 Feb 18;76(4):720-729. doi: 10.1093/cid/ciac130. PMID 35235656
- [Derived] Kumar P, Clarke AE, Jonsson-Oldenbuttel C, Deltoro MG, Di Giambenedetto S, Brites C, Hocqueloux L, Lu PL, Oyee J, Oglesby A, Wynne B, Jones B, Evitt LA, Fox D, Kisare M, Priest J. Patient-Reported Outcomes After Switching to a 2-Drug Regimen of Fixed-Dose Combination Dolutegravir/Lamivudine: 48-Week Results from the SALSA Study. AIDS Behav. 2025 Jan;29(1):235-245. doi: 10.1007/s10461-024-04479-9. Epub 2024 Sep 3. PMID 39225890
- [Derived] Scholten S, Cahn P, Portilla J, Bisshop F, Hodder S, Ruane P, Kaplan R, Wynne BR, Man CY, Grove R, Wang R, Jones B, Ait-Khaled M, Kisare M, Okoli C. Dolutegravir/Lamivudine Efficacy and Safety Outcomes in People With HIV-1 With or Without Historical Resistance Results at Screening: 48-Week Pooled Analysis. Open Forum Infect Dis. 2024 Jul 1;11(7):ofae365. doi: 10.1093/ofid/ofae365. eCollection 2024 Jul. PMID 39015350
- [Derived] Walmsley S, Smith DE, Gorgolas M, Cahn PE, Lutz T, Lacombe K, Kumar PN, Wynne B, Grove R, Bontempo G, Moodley R, Okoli C, Kisare M, Jones B, Clark A, Ait-Khaled M. Efficacy and safety of switching to dolutegravir/lamivudine in virologically suppressed people with HIV-1 aged >/= 50 years: week 48 pooled results from the TANGO and SALSA studies. AIDS Res Ther. 2024 Mar 21;21(1):17. doi: 10.1186/s12981-024-00604-9. PMID 38515183
- [Derived] Masters MC, Cohn SE. Two-drug HIV regimens: more data still needed. Lancet HIV. 2021 Aug;8(8):e454-e455. doi: 10.1016/S2352-3018(21)00106-5. No abstract available. PMID 34358493

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consist of two phases - Randomized phase and Continuation phase.
Pre-assignment Details: A total of 493 adult participants were enrolled in this study. Continuation Phase was not applicable for participants in Sweden and Denmark.
Groups:
- Randomized Phase-Participants Who Received DTG/3TC FDC: Eligible participants were randomized to receive 50 milligrams (mg)/300 mg DTG/3TC FDC therapy from day 1 up to 52 weeks. Participants who completed 52 weeks of treatment had the opportunity to continue receiving DTG/3TC FDC once daily in the continuation phase.
- Randomized Phase-Participants Who Received CAR: Eligible participants received CAR from day 1 up to 52 weeks. CAR included 2 nucleoside reverse transcriptase inhibitors (NTRIs) plus either an integrase inhibitor (INI), non-nucleoside reverse transcriptase inhibitor (NNRTI), or boosted protease inhibitor (PI) or atazanavir unboosted.
- Continuation Phase-Participants Who Received DTG/3TC FDC: Participants who completed 52 weeks of treatment of DTG/3TC FDC had the opportunity to continue receiving DTG/3TC FDC once daily in the continuation phase up to week 132.
Period: Randomized Phase (Day1 to Week 52)
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR | Continuation Phase-Participants Who Received DTG/3TC FDC
Started | 246 | 247 | 0
Completed | 136 | 229 | 0
Not Completed | 110 | 18 | 0
Not completed — Adverse Event | 4 | 3 | 0
Not completed — Lack of Efficacy | 0 | 3 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Physician Decision | 1 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 5 | 0
Not completed — Transferred to continuation phase | 96 | 0 | 0
Not completed — Protocol Deviation | 5 | 4 | 0
Period: Continuation Phase (Week 52 to Week 132)
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR | Continuation Phase-Participants Who Received DTG/3TC FDC
Started | 0 (This consist of participants who got transferred to continuation phase.) | 0 (Participants did not receive CAR in continuation phase.) | 96 (Transferred to continuation phase)
Completed | 0 | 0 | 91
Not Completed | 0 | 0 | 5
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR | Total
Number analyzed (Participants) | 246 | 247 | 493
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 45.5 (11.04) | 45.8 (11.99) | 45.7 (11.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 84 | 192
  Male | 138 | 163 | 301
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 45 | 48 | 93
  American Indian OR Alaska Native | 18 | 14 | 32
  Asian - East Asian Heritage | 27 | 36 | 63
  Asian - South East Asian Heritage | 4 | 3 | 7
  White - Arabic/North African Heritage | 7 | 4 | 11
  White - White/Caucasian/European Heritage | 142 | 140 | 282
  Multiple | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Plasma HIV-1 Ribonucleic Acid (RNA) >=50 Copies/Milliliter (c/mL) as Per Food and Drug Administration (FDA) Snapshot Category at Week 48
Description: Number of participants with plasma HIV 1 RNA >=50 c/mL were evaluated using FDA snapshot algorithm at Week 48 to demonstrate the non-inferior antiviral activity of switching to DTG/3TC FDC once daily compared to continuation of CAR over 48 weeks. The FDA snapshot algorithm defines a participant's virologic response status using only the viral load at the predefined time point within a window of time (HIV-RNA equal to or above 50 copies/mL and HIV-RNA below 50 copies/mL ), along with study drug discontinuation status. Participants with plasma HIV 1 RNA >=50 c/mL were termed as subjects with virologic failure. The third category of the FDA snapshot ("No virologic data") is not pre-defined as an endpoint and therefore not reported separately.
Time Frame: Week 48
Population: Intent To Treat-Exposed (ITT-E) population included all randomized participants who received at least one dose of study medication either DTG/3TC or CAR.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 246 | 247
Participants | 1 | 3
Statistical Analysis 1: Comparison: Randomized Phase-Participants Who Received DTG/3TC FDC vs Randomized Phase-Participants Who Received CAR; Test type: Non-Inferiority — Non-inferiority was be concluded if the upper bound of the two-sided 95% confidence interval (CI) for the CMH adjusted difference in the proportion of patients with plasma HIV-1 RNA ≥ 50 c/mL between each treatment group (DTG/3TC - CAR) is less than 5%; Adjusted Difference in Percent (ADP) = -0.8, 95% CI 2-sided [-2.4 to 0.8] — ADP was based on Cochran-Mantel Haenszel stratified analysis adjusting for Baseline stratification factor:Baseline third agent (protease inhibitor [PI], non-nucleoside reverse transcriptase inhibitor [NNRTI], and integrase inhibitor [INI])

2. Secondary Outcome: Number of Participants With Plasma HIV-1 RNA <50 c/mL Using the FDA Snapshot Algorithm at Week 48
Description: Number of participants with plasma HIV 1 RNA <50 c/mL were evaluated using FDA snapshot algorithm at Week 48 to demonstrate the antiviral activity of switching to DTG/3TC FDC once daily compared to continuation of CAR over 48 weeks. The FDA snapshot algorithm defines a participant's virologic response status using only the viral load at the predefined time point within a window of time (HIV-RNA equal to or above 50 copies/mL and HIV-RNA below 50 copies/mL ), along with study drug discontinuation status. Participants with plasma HIV 1 RNA <50 c/mL were termed as subjects with virologic success. The third category of the FDA snapshot ("No virologic data") is not pre-defined as an endpoint and therefore not reported separately.
Time Frame: Week 48
Population: Intent To Treat-Exposed
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 246 | 247
Participants | 232 | 229
Statistical Analysis 1: Comparison: Randomized Phase-Participants Who Received DTG/3TC FDC vs Randomized Phase-Participants Who Received CAR; Test type: Non-Inferiority — Non-inferiority will be concluded if the lower bound of a 2-sided 95% confidence interval for the difference in success rates between the two treatment arms (DTG/3TC-CAR) is greater than -12%; Adjusted Difference in Percent = 1.6, 95% CI 2-sided [-2.8 to 5.9] — ADP was based on Cochran-Mantel Haenszel stratified analysis adjusting for Baseline stratification factor:Baseline third agent (PI, NNRTI, and INI)

3. Secondary Outcome: Number of Participants With Plasma HIV-1 RNA >=50 c/mL as Per FDA Snapshot Category at Week 24
Description: Number of participants with plasma HIV 1 RNA >=50 c/mL were evaluated using FDA snapshot algorithm at Week 24 to demonstrate the antiviral activity of switching to DTG/3TC FDC once daily compared to continuation of CAR over 24 weeks. The FDA snapshot algorithm defines a participant's virologic response status using only the viral load at the predefined time point within a window of time (HIV-RNA equal to or above 50 copies/mL and HIV-RNA below 50 copies/mL ), along with study drug discontinuation status. Participants with plasma HIV 1 RNA >=50 c/mL were termed as subjects with virologic failure. The third category of the FDA snapshot ("No virologic data") is not pre-defined as an endpoint and therefore not reported separately.
Time Frame: Week 24
Population: Intent To Treat-Exposed
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 246 | 247
Participants | 0 | 1

4. Secondary Outcome: Number of Participants With Plasma HIV-1 RNA <50 c/mL Using the FDA Snapshot Algorithm at Week 24
Description: Number of participants with plasma HIV 1 RNA <50 c/mL were evaluated using FDA snapshot algorithm at Week 24 to demonstrate the antiviral activity of switching to DTG/3TC FDC once daily compared to continuation of CAR over 24 weeks. The FDA snapshot algorithm defines a participant's virologic response status using only the viral load at the predefined time point within a window of time (HIV-RNA equal to or above 50 copies/mL and HIV-RNA below 50 copies/mL ), along with study drug discontinuation status. Participants with plasma HIV 1 RNA <50 c/mL were termed as subjects with virologic success. The third category of the FDA snapshot ("No virologic data") is not pre-defined as an endpoint and therefore not reported separately.
Time Frame: Week 24
Population: Intent To Treat-Exposed
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 246 | 247
Participants | 234 | 237

5. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4 (CD4+) Cell Count for Week 24
Description: CD4+ cells are type of white blood cells that fight infection and as HIV infection progresses, the number of these cells declines. Baseline value is defined as the latest pre-dose assessment with a non-missing value (Day 1). Change from Baseline is defined as post-dose visit value minus Baseline value. Lymphocyte subsets were collected for assessment of this outcome measure by flow cytometry. Change from Baseline in CD4+ lymphocyte count was assessed at Week 24 to evaluate the immune effects of DTG/3TC FDC once daily compared to continuation of CAR. Plasma samples for lymphocyte subsets were collected.
Time Frame: Baseline (Day 1) and Week 24
Population: Intent To Treat-Exposed. Only those participants with data available at specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: cells/cubic millimeter (cells/mm^3)
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 232 | 235
cells/cubic millimeter (cells/mm^3) | 30.5 [-71.5 to 111] | 10 [-79 to 95]

6. Secondary Outcome: Change From Baseline in CD4+ Cell Count for Week 48
Description: CD4+ cells are type of white blood cells that fight infection and as HIV infection progresses, the number of these cells declines. Baseline value is defined as the latest pre-dose assessment with a non-missing value (Day 1). Change from Baseline is defined as post-dose visit value minus Baseline value. Lymphocyte subsets were collected for assessment of this outcome measure by flow cytometry. Change from Baseline in CD4+ lymphocyte count was assessed at Week 48 to evaluate the immune effects of DTG/3TC FDC once daily compared to continuation of CAR. Plasma samples for lymphocyte subsets were collected.
Time Frame: Baseline (Day 1) and Week 48
Population: Intent To Treat-Exposed. Only those participants with data available at specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 232 | 227
cells/mm^3 | 30 [-83 to 115.5] | 2 [-105 to 94]

7. Secondary Outcome: Change From Baseline in CD4+/ Cluster of Differentiation 8 (CD8+) Cell Counts Ratio for Week 24
Description: CD4+/CD8+ cells are type of white blood cells that fight infection and as HIV infection progresses, the number of these cells declines. Baseline value is defined as the latest pre-dose assessment with a non-missing value (Day 1). Change from Baseline is defined as post-dose visit value minus Baseline value. Lymphocyte subsets were collected for assessment of this outcome measure by flow cytometry. Change from Baseline in CD4+/CD8+ lymphocyte cell count ratio was assessed at Week 24 to evaluate the immune effects of DTG/3TC FDC once daily compared to continuation of CAR. Plasma samples for lymphocyte subsets were collected.
Time Frame: Baseline (Day 1) and Week 24
Population: Intent To Treat-Exposed. Only those participants with data available at specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 232 | 235
Ratio | -0.02 [-0.105 to 0.07] | 0.01 [-0.06 to 0.09]

8. Secondary Outcome: Change From Baseline in CD4+/CD8+ Cell Counts Ratio for Week 48
Description: CD4+/CD8+ cells are type of white blood cells that fight infection and as HIV infection progresses, the number of these cells declines. Baseline value is defined as the latest pre-dose assessment with a non-missing value (Day 1). Change from Baseline is defined as post-dose visit value minus Baseline value. Lymphocyte subsets were collected for assessment of this outcome measure by flow cytometry. Change from Baseline in CD4+/CD8+ lymphocyte cell count ratio was assessed at Week 48 to evaluate the immune effects of DTG/3TC FDC once daily compared to continuation of CAR. Plasma samples for lymphocyte subsets were collected.
Time Frame: Baseline (Day 1) and Week 48
Population: Intent To Treat-Exposed. Only those participants with data available at specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 232 | 227
Ratio | 0.04 [-0.06 to 0.13] | 0.05 [-0.06 to 0.13]

9. Secondary Outcome: Number of Participants With Disease Progression Through Week 24
Description: Participants with disease progression included incidences of HIV-associated conditions, Acquired Immuno Deficiency Syndrome (AIDS) and death. HIV-associated conditions were assessed according to the 2014 HIV infection by Centers for Disease Control and Prevention (CDC) classification system for HIV Infection in adults to evaluate the immune effects of DTG /3TC FDC once daily compared to continuation of CAR.
Time Frame: Up to Week 24
Population: Intent To Treat-Exposed
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 246 | 247
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With Disease Progression Through Week 48
Description: Participants with disease progression included incidences of HIV-associated conditions, AIDS and death. HIV-associated conditions were assessed according to the 2014 HIV infection by CDC classification system for HIV Infection in adults to evaluate the immune effects of DTG /3TC FDC once daily compared to continuation of CAR.
Time Frame: Up to Week 48
Population: Intent To Treat-Exposed
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 246 | 247
Participants | 1 | 0

11. Secondary Outcome: Number of Participants With Adverse Events (AEs) and AEs Leading to Discontinuation
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Time Frame: Up to Week 52
Population: Safety population included all randomized participants who received at least 1 dose of study intervention either DTG/3TC or CAR.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 246 | 247
Participants
  AEs | 180 | 172
  AEs leading to discontinuation | 5 | 3

12. Secondary Outcome: Number of Participants With AEs by Severity Grades
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs were evaluated by the investigator and graded according to the Division of Acquired Immunodeficiency Syndrome (DAIDS) toxicity scales from Grade 1 to 5 (1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening, 5=Death). The higher the grade, the more severe the symptoms
Time Frame: Up to 52 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 246 | 247
Participants
  Grade 1 | 92 | 67
  Grade 2 | 77 | 86
  Grade 3 | 10 | 17
  Grade 4 | 0 | 2
  Grade 5 | 1 | 0

13. Secondary Outcome: Number of Participants With Hepatobiliary Abnormalities Through 52 Weeks
Description: Blood samples were collected to evaluate hepatobiliary abnormalities. Number of participants with Bilirubin (BIL), Alkaline phosphatase (ALP), Alanine Aminotransferase (ALT)/combination of these with levels more than the defined hepatobiliary abnormality criteria were presented. Hepatocellular injury is defined as ([ALT/ALT ULN]/[ALP/ALP ULN]) >= 5 and ALT >=3xULN.
Time Frame: Up to Week 52
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 246 | 247
Participants
  ALT >=3xUpper Limit of Normal (ULN) & BIL >=2xULN | 0 | 0
  ALT >=3xULN & ALP <2xULN & BIL >=2xULN | 0 | 0
  ALT >=3xULN & BIL >=1.5xULN | 0 | 0
  AST >=3xULN & BIL >=2xULN | 0 | 0
  AST >=3xULN & ALP <2xULN & BIL >=2xULN | 0 | 0
  AST >=3xULN & BIL >=1.5xULN | 0 | 0
  ALT+AST >=20xULN | 0 | 0
  ALT+AST >=10xULN | 0 | 0
  ALT+AST >=5xULN | 0 | 0
  ALT+AST >=3xULN | 3 | 2
  ALT >=20xULN | 0 | 0
  ALT >=10xULN | 0 | 0
  ALT >=5xULN | 1 | 1
  ALT >=3xULN | 6 | 5
  AST >=20xULN | 0 | 0
  AST >=10xULN | 0 | 0
  AST >=5xULN | 1 | 0
  AST >=3xULN | 5 | 2
  BIL >=2xULN | 0 | 5
  BIL >=1.5xULN | 0 | 7
  ALP >=1.5xULN | 4 | 8
  ALT >=3xULN - <5xULN | 5 | 4
  ALT >=5xULN - <10xULN | 1 | 1
  ALT >=10xULN - <20xULN | 0 | 0
  Hepatocellular injury | 5 | 1
  Hepatocellular injury and BIL >=2xULN | 0 | 0

14. Secondary Outcome: Number of Participants With Any AEs and AEs by Severity Grades for Those Participants With Baseline Creatinine Clearance of 30-49 mL/Min/1.73m^2
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Number of participants with any AE were presented and AEs were graded according to the DAIDS toxicity scales from Grade 1 to 5 (1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening, 5=Death). The higher the grade, the more severe the symptoms.
Time Frame: Up to 52 weeks
Population: Safety population. Only those participants with data available at specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 1 | 4
Participants
  Any Event | 1 | 3
  Grade 1 | 1 | 1
  Grade 2 | 0 | 2
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

15. Secondary Outcome: Number of Participants With Any AEs and AEs by Severity Grades for Those Participants With Baseline Creatinine Clearance of >=50 mL/Min/1.73m^2
Description: as for outcome 14
Time Frame: Up to 52 weeks
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 245 | 243
Participants
  Any Event | 179 | 169
  Grade 1 | 91 | 66
  Grade 2 | 77 | 84
  Grade 3 | 10 | 17
  Grade 4 | 0 | 2
  Grade 5 | 1 | 0

16. Secondary Outcome: Number of Participants With Any AEs Leading to Discontinuation Based on Baseline Creatinine Clearance of 30-49 mL/Min/1.73m^2
Description: as for outcome 11
Time Frame: Up to 52 weeks
Population: Safety population. Only those participants with data available at specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 1 | 4
Participants | 0 | 1

17. Secondary Outcome: Number of Participants With Any AEs Leading to Discontinuation Based on Baseline Creatinine Clearance of >=50 mL/Min/1.73m^2
Description: as for outcome 11
Time Frame: Up to 52 weeks
Population: Safety population. Only those participants with data available at specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 245 | 243
Participants | 5 | 2

18. Secondary Outcome: Number of Participants With Hepatobiliary Abnormalities Through 52 Weeks Based on Baseline Creatinine Clearance of 30-49 mL/Min/1.73m^2
Description: as for outcome 13
Time Frame: Up to Week 52
Population: Safety population. Only those participants with data available at specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 1 | 4
Participants
  ALT >=3xUpper Limit of Normal (ULN) & BIL >=2xULN | 0 | 0
  ALT >=3xULN & ALP <2xULN & BIL >=2xULN | 0 | 0
  ALT >=3xULN & BIL >=1.5xULN | 0 | 0
  AST >=3xULN & BIL >=2xULN | 0 | 0
  AST >=3xULN & ALP <2xULN & BIL >=2xULN | 0 | 0
  AST >=3xULN & BIL >=1.5xULN | 0 | 0
  ALT+AST >=20xULN | 0 | 0
  ALT+AST >=10xULN | 0 | 0
  ALT+AST >=5xULN | 0 | 0
  ALT+AST >=3xULN | 0 | 0
  ALT >=20xULN | 0 | 0
  ALT >=10xULN | 0 | 0
  ALT >=5xULN | 0 | 0
  ALT >=3xULN | 0 | 0
  AST >=20xULN | 0 | 0
  AST >=10xULN | 0 | 0
  AST >=5xULN | 0 | 0
  AST >=3xULN | 0 | 0
  BIL >=2xULN | 0 | 1
  BIL >=1.5xULN | 0 | 1
  ALP >=1.5xULN | 0 | 0
  ALT >=3xULN - <5xULN | 0 | 0
  ALT >=5xULN - <10xULN | 0 | 0
  ALT >=10xULN - <20xULN | 0 | 0
  Hepatocellular injury | 0 | 0
  Hepatocellular injury and BIL >=2xULN | 0 | 0

19. Secondary Outcome: Number of Participants With Hepatobiliary Abnormalities Through 52 Weeks Based on Baseline Creatinine Clearance of >=50 mL/Min/1.73m^2
Description: as for outcome 13
Time Frame: Up to Week 52
Population: Safety population. Only those participants with data available at specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 245 | 243
Participants
  ALT >=3xUpper Limit of Normal (ULN) & BIL >=2xULN | 0 | 0
  ALT >=3xULN & ALP <2xULN & BIL >=2xULN | 0 | 0
  ALT >=3xULN & BIL >=1.5xULN | 0 | 0
  AST >=3xULN & BIL >=2xULN | 0 | 0
  AST >=3xULN & ALP <2xULN & BIL >=2xULN | 0 | 0
  AST >=3xULN & BIL >=1.5xULN | 0 | 0
  ALT+AST >=20xULN | 0 | 0
  ALT+AST >=10xULN | 0 | 0
  ALT+AST >=5xULN | 0 | 0
  ALT+AST >=3xULN | 3 | 2
  ALT >=20xULN | 0 | 0
  ALT >=10xULN | 0 | 0
  ALT >=5xULN | 1 | 1
  ALT >=3xULN | 6 | 5
  AST >=20xULN | 0 | 0
  AST >=10xULN | 0 | 0
  AST >=5xULN | 1 | 0
  AST >=3xULN | 5 | 2
  BIL >=2xULN | 0 | 4
  BIL >=1.5xULN | 0 | 6
  ALP >=1.5xULN | 4 | 8
  ALT >=3xULN - <5xULN | 5 | 4
  ALT >=5xULN - <10xULN | 1 | 1
  ALT >=10xULN - <20xULN | 0 | 0
  Hepatocellular injury | 5 | 1
  Hepatocellular injury and BIL >=2xULN | 0 | 0

20. Secondary Outcome: Change From Baseline in Fasting Lipids at Week 24
Description: Lipid parameters included total cholesterol, high density lipoprotein (HDL) cholesterol, low density lipoprotein (LDL) cholesterol and triglycerides.
Time Frame: Baseline (Day 1) and Week 24
Population: Safety Population. Only those participants with data available at specified time points has been analyzed.
Measure: Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 191 | 168
milligram/deciliter (mg/dL)
  Serum or Plasma Triglycerides (mg/dL) | -4.944 (56.4947) | -3.571 (61.9494)
  Serum or Plasma HDL Cholesterol, Direct (mg/dL) | -0.326 (9.1737) | 0.585 (8.3277)
  Serum or Plasma Cholesterol (mg/dL) | -3.096 (31.6634) | 0.058 (25.8019)
  Serum or Plasma LDL Cholesterol (Calculated or Direct), (mg/dL) | -1.64 (25.5153) | -0.06 (19.802)

21. Secondary Outcome: Change From Baseline in Fasting Lipids at Week 48
Description: Lipid parameters included total cholesterol, HDL cholesterol, LDL cholesterol and triglycerides.
Time Frame: Baseline (Day 1) and Week 48
Population: Safety Population. Only those participants with data available at specified time points has been analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 186 | 159
mg/dL
  Serum or Plasma Triglycerides (mg/dL) | -3.112 (66.9065) | -4.002 (71.0132)
  Serum or Plasma HDL Cholesterol, Direct (mg/dL) | -0.809 (10.5651) | 0.688 (8.5584)
  Serum or Plasma Cholesterol (mg/dL) | 0.131 (30.271) | 2.668 (27.0351)
  Serum or Plasma LDL Cholesterol (Calculated or Direct), (mg/dL) | 1.753 (22.8585) | 2.734 (20.0256)

22. Secondary Outcome: Number of Participants With Observed Genotypic and Phenotypic Resistance to Antiretrovirals (ARVs) for Participants Meeting Confirmed Virologic Withdrawal (CVW) Criteria
Description: Genotypic and phenotypic testing was conducted for participants who met the CVW criteria, i.e., one assessment with HIV-1 RNA ≥200 c/mL after Day 1 with an immediately prior HIV-1 RNA ≥50 c/mL at any point in the study.
Time Frame: Up to week 48
Population: Confirmed Virologic Withdrawal (CVW) population. No participants met the CVW criteria over 48 weeks; therefore, the genotypic and phenotypic resistance virologic analyses were not assessed.
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Change From Baseline in Health Status by HIV Treatment Satisfaction Questionnaire (TSQ) at Week 24
Description: The HIV Treatment Satisfaction Questionnaire (HIVTSQ) is a 10-item self-reported scale that consists of a total score ranging from 0 to 60. Higher scores indicate a greater level of patient-reported satisfaction with their current therapy.
Time Frame: Baseline (Day 1) and Week 24
Population: ITT-E. Only those participants with data available at specified time points has been analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 236 | 240
Scores on a scale | 2.9 (5.85) | 1 (5.16)
Statistical Analysis 1: Comparison: Randomized Phase-Participants Who Received DTG/3TC FDC vs Randomized Phase-Participants Who Received CAR; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Adjusted Mean = 1.4, 95% CI 2-sided [0.7 to 2.2] — MMRM adjusted for following: Treatment, Visit, Baseline Third Agent Class, Age (continuous), Sex, Race, Baseline Value (continuous), Treatment by Visit interaction, Baseline Value by Visit interaction, with Visit as the repeated factor

24. Secondary Outcome: Change From Baseline in Health Status by HIV TSQ at Week 48
Description: The HIVTSQ is a 10-item self-reported scale that consists of a total score ranging from 0 to 60. Higher scores indicate a greater level of patient-reported satisfaction with their current therapy.
Time Frame: Baseline (Day 1) and Week 48
Population: ITT-E. Only those participants with data available at specified time points has been analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 229 | 229
Scores on a scale | 2.9 (6) | 1 (5.14)
Statistical Analysis 1: Comparison: Randomized Phase-Participants Who Received DTG/3TC FDC vs Randomized Phase-Participants Who Received CAR; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Adjusted Mean = 1.4, 95% CI 2-sided [0.7 to 2.2] — [estimate comment as in outcome 23, analysis 1]

25. Secondary Outcome: Change From Baseline in Health Status by Symptom Distress Module (SDM) at Week 24
Description: SDM is a 20-item self-reported measure that addresses the presence and perceived distress linked to symptoms commonly associated with HIV or its treatment. Each item is rated from 0 to 4 where 0 (complete absence of symptom) and 4 (very bothersome symptom). Overall score calculated as the sum of the scores for each of the 20 items of the questionnaire and ranged from 0 (best health) and 80 (worst health).
Time Frame: Baseline (Day 1) and Week 24
Population: ITT-E. Only those participants with data available at specified time points has been analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 235 | 239
Scores on a scale | -2.6 (8.69) | -0.7 (8.01)
Statistical Analysis 1: Comparison: Randomized Phase-Participants Who Received DTG/3TC FDC vs Randomized Phase-Participants Who Received CAR; Test type: Other; p = 0.021, Mixed Model Repeated Measures; Adjusted Mean = -1.6, 95% CI 2-sided [-2.9 to -0.2] — [estimate comment as in outcome 23, analysis 1]

26. Secondary Outcome: Change From Baseline in Health Status by SDM at Week 48
Description: as for outcome 25
Time Frame: Baseline (Day 1) and Week 48
Population: ITT-E. Only those participants with data available at specified time points has been analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR
Number analyzed (Participants) | 228 | 226
Scores on a scale | -2.4 (7.64) | -1.5 (7.92)
Statistical Analysis 1: Comparison: Randomized Phase-Participants Who Received DTG/3TC FDC vs Randomized Phase-Participants Who Received CAR; Test type: Other; p = 0.398, Mixed Model Repeated Measures; Adjusted Mean = -0.5, 95% CI 2-sided [-1.8 to 0.7] — [estimate comment as in outcome 23, analysis 1]

27. Secondary Outcome: Change From Baseline in Health Status by SDM in Continuation Phase
Description: as for outcome 25
Time Frame: Baseline (Day 1) and Week 76, Week 100, and Week 132
Population: Intent To Treat-Exposed (ITT-E) Continuation Phase population included participants who received at least one dose of DTG/3TC during continuation phase. Only those participants with data available at specified time points has been analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Continuation Phase-Participants Who Received DTG/3TC FDC
Number analyzed (Participants) | 96
Scores on a scale
  Week 76: number analyzed (Participants) | 56
  Week 76 | -4.1 (8.69)
  Week 100: number analyzed (Participants) | 26
  Week 100 | -3.4 (11.33)
  Week 132: number analyzed (Participants) | 32
  Week 132 | -6.1 (9.94)

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious adverse events (non-SAEs) and serious adverse events (SAEs) were collected from day 1 to week 52 for Randomized Phase and from week 52 to week 132 for continuation phase.
Description: Safety Population included all randomized participants who received at least 1 dose of study intervention.
Arm/Group | Randomized Phase-Participants Who Received DTG/3TC FDC | Randomized Phase-Participants Who Received CAR | Continuation Phase-Participants Who Received DTG/3TC FDC
All-Cause Mortality (participants affected / at risk) | 1/246 | 0/247 | 0/96
Serious Adverse Events (participants affected / at risk) | 7/246 | 16/247 | 1/96
Other Adverse Events (participants affected / at risk) | 179/246 | 169/247 | 43/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Phase-Participants Who Received DTG/3TC FDC (N=246) | Randomized Phase-Participants Who Received CAR (N=247) | Continuation Phase-Participants Who Received DTG/3TC FDC (N=96)
COVID-19 (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Phase-Participants Who Received DTG/3TC FDC (N=246) | Randomized Phase-Participants Who Received CAR (N=247) | Continuation Phase-Participants Who Received DTG/3TC FDC (N=96)
Headache (Nervous system disorders) | 16 (18) | 17 (20) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 11 (11) | 15 (16) | 3 (3)
Weight increased (Investigations) | 20 (20) | 5 (5) | 3 (3)
COVID-19 (Infections and infestations) | 14 (14) | 8 (8) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (15) | 7 (7) | 3 (3)
Nasopharyngitis (Infections and infestations) | 11 (12) | 9 (10) | 3 (3)
Dizziness (Nervous system disorders) | 13 (15) | 6 (7) | 1 (1)
Insomnia (Psychiatric disorders) | 14 (15) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 10 (11) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 8 (9) | 0 (0)
Syphilis (Infections and infestations) | 9 (10) | 5 (5) | 1 (1)
Hypertension (Vascular disorders) | 6 (7) | 7 (7) | 2 (2)
Pyrexia (General disorders) | 6 (8) | 7 (7) | 0 (0)
Anxiety (Psychiatric disorders) | 5 (5) | 6 (6) | 5 (5)
Fatigue (General disorders) | 5 (5) | 6 (6) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 7 (7) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (7) | 4 (6) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 5 (7) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3) | 5 (5) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (6) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (4) | 5 (5) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 5 (6) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 6 (6) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 6 (7) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 4 (4) | 3 (3) | 0 (0)
Blood creatinine increased (Investigations) | 3 (3) | 3 (3) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 5 (5)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 5 (5)
Low density lipoprotein increased (Investigations) | 2 (2) | 4 (4) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 1 (1)
Sleep disorder (Psychiatric disorders) | 3 (3) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 2 (3) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 1 (1)
Blood cholesterol increased (Investigations) | 2 (2) | 3 (3) | 2 (2)
Conjunctivitis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 4 (4) | 1 (1)
Toothache (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 3 (3) | 0 (0)
Chlamydial infection (Infections and infestations) | 2 (2) | 2 (3) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 0 (0)
Onychomycosis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Proctitis gonococcal (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 2 (2) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 2 (2)
Dental caries (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 1 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 1 (1) | 0 (0)
Insulin resistance (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Oropharyngeal gonococcal infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 1 (2) | 2 (2)
Blood triglycerides increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Creatinine renal clearance increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 2 (2) | 0 (0) | 3 (3)
Gonococcal infection (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Gonorrhoea (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Loss of libido (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Metabolic syndrome (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Primary syphilis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Sensory loss (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Urine protein/creatinine ratio increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acromegaly (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Anal chlamydia infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anogenital dysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anorectal human papilloma virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anosmia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Blood glucose abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood insulin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood prolactin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 1 (1) | 0 (0)
Body tinea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bone formation increased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Crystal urine present (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dental restoration failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes insipidus (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dysplastic naevus syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Essential hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Finger deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastric cyst (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric dilatation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Genital herpes simplex (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Genitourinary chlamydia infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Glucose urine present (Investigations) | 0 (0) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hemianopia heteronymous (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Initial insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Lichen planus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Menstruation delayed (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Neck injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Ocular hypertension (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (2) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic organ injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Penis injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (3) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal chlamydia infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 1 (1) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pseudofolliculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pulse absent (Investigations) | 0 (0) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Secondary hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Secondary syphilis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin plaque (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Solar lentigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Stress at work (Social circumstances) | 0 (0) | 1 (1) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroid disorder (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Tinea capitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urethritis gonococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urine albumin/creatinine ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vasodilatation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bell's palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lymph gland infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Device physical property issue (Product Issues) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/90/NCT04021290/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/90/NCT04021290/SAP_002.pdf